CLINICAL TRIAL: NCT01653821
Title: Surgical Removal of Carotid Body in Patients With Systolic Heart Failure.
Acronym: FIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Noblewell (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIM-WROCPL-CORIDEA
Record Dates: First submitted 2012-07-26; First posted 2012-07-31 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Systolic Heart Failure; Peripheral Chemoreceptor Hypersensitivity
Keywords: carotid body; heart failure; chemoreceptor; hypersensitivity
MeSH Terms: conditions — Heart Failure, Systolic; Heart Failure; Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Carotid body excision (Experimental): Patients undergoing unilateral or bilateral removal of carotid body.
  Interventions: Procedure: Carotid body excision

INTERVENTIONS:
Procedure: Carotid body excision

SUMMARY:
The aim of the study is to determine safety, tolerability and feasibility of unilateral and bilateral carotid body excision in patients with systolic heart failure and peripheral chemoreceptor hypersensitivity.

ELIGIBILITY:
Inclusion Criteria:

* History of heart failure class II-III according to NYHA within at least 6 months prior to inclusion
* Stable clinical state within at least 4 weeks prior to inclusion
* Subject >= 18 years old
* Left ventricular ejection fraction ≤ 45% evaluated by transthoracic echocardiography (Simpson's method)
* Carotid body present in computer cervical angiotomography
* History of exacerbated peripheral chemoreceptor sensitivity determined as >0.6L/min/%SpO2
* Able and willing to give written informed consent

Exclusion Criteria:

* Unstable angina pectoris, coronary attack, coronary revascularization, exacerbation of heart-failure requiring hospitalization, clinically significant infection, surgery under general anesthesia within 3 months prior to inclusion
* History of stroke, transient ischemic attack (TIA), or clinically significant chronic neurological disorder
* History of heart transplant
* Pregnancy or anticipation of pregnancy
* Hemodialysis or peritoneal dialysis patients
* Obstructive carotid atherosclerotic disease with >50% stenosis
* Severe sleep apnea syndrome diagnosed in PSG
* COPD stage III and IV according to GOLD 2007
* Unable to perform the spiroergometric assessment
* Any significant anomaly in additional investigation which may increase the risk of study procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Peripheral chemosensitivity | 4 weeks
  Ventilatory response to hypoxia using transient inhalation of nitrogen.

CONTACTS AND LOCATIONS:
Locations (1):
- Centrum Chorób Serca - Klinika Kardiologii, 4. Wojskowy Szpital Kliniczny, Wroclaw, Poland

REFERENCES:
- [Derived] Niewinski P, Janczak D, Rucinski A, Jazwiec P, Sobotka PA, Engelman ZJ, Fudim M, Tubek S, Jankowska EA, Banasiak W, Hart EC, Paton JF, Ponikowski P. Carotid body removal for treatment of chronic systolic heart failure. Int J Cardiol. 2013 Oct 3;168(3):2506-9. doi: 10.1016/j.ijcard.2013.03.011. Epub 2013 Mar 29. PMID 23541331